CLINICAL TRIAL: NCT01014975
Title: A Phase 1/2a, Open Label, Dose Escalation, Safety Study of Intra-thrombus Plasmin (Human) Administration in Acute, Middle Cerebral Artery, Ischemic Stroke
Brief Title: A Safety and Dose Finding Study of Plasmin (Human) Administered Into the Middle Cerebral Artery of Stroke Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T05018-1001; 2010-019760-36 (EudraCT Number)
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Acute Ischemic Stroke
Keywords: stroke; plasmin; thrombus; ischemic; middle cerebral artery; thrombolysis; intra-arterial; fibrin
MeSH Terms: conditions — Ischemic Stroke; Stroke; Thrombosis; Ischemia | interventions — Fibrinolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 20 mg Plasmin (Human) (Experimental): 20 mg of Plasmin (Human)
  Interventions: Biological: Plasmin (Human)
- 40 mg Plasmin (Human) (Experimental): 40 mg of Plasmin (Human)
  Interventions: Biological: Plasmin (Human)
- 80 mg Plasmin (Human) (Experimental): 80 mg of Plasmin (Human)
  Interventions: Biological: Plasmin (Human)

INTERVENTIONS:
Biological: Plasmin (Human) — Plasmin (Human), 20 mg, delivered through a catheter into a thrombus
  Other Names: TAL-05-00018; BAY-57-9602
  Arms: 20 mg Plasmin (Human)
Biological: Plasmin (Human) — Plasmin (Human), 40 mg, delivered through a catheter into a thrombus
  Other Names: TAL-05-00018; BAY-57-9602
  Arms: 40 mg Plasmin (Human)
Biological: Plasmin (Human) — Plasmin (Human), 80 mg, delivered through a catheter into a thrombus
  Other Names: TAL-05-00018; BAY-57-9602
  Arms: 80 mg Plasmin (Human)

SUMMARY:
This study tests the drug, Plasmin (Human), in patients with a stroke due to a clot in the middle cerebral artery (MCA). Plasmin is an enzyme that causes clot lysis by cleaving a clot component, fibrin. In this study, Plasmin (Human) is administered locally through a catheter to the clot within 9 hours of the stroke onset. Three doses of Plasmin (Human) (20 mg, 40 mg, and 80 mg) are being tested in 3 different groups of patients. Patients are monitored by imaging of the affected artery and functional testing.

DETAILED DESCRIPTION:
This is a Phase 1/2a, open-label, multi-center, sequential dose escalation, safety study of Plasmin (Human) in acute ischemic stroke caused by middle cerebral artery occlusion documented by arteriography. Plasmin (Human) will be administered through a catheter into the thrombus within 9 hours of stroke onset. Approximately sixty-one (61) patients will be enrolled and will receive Plasmin (Human). The objectives of this study are to determine the safety of escalating doses of Plasmin (Human) and to determine the proportion of patients with treatment success, defined as partial or full recanalization.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 85 years of age
2. Male or female
3. New focal, potentially disabling neurologic deficit clinically localized to the MCA distribution
4. Intra-arterial therapy with Plasmin completed within 9 hours of stroke onset
5. A National Institutes of Health Stroke Scale score ≥ 4 and ≤ 25

Exclusion Criteria:

1. Intracranial procedures or intracranial or systemic bleeding within the last year
2. Intracranial neoplasm (except meningioma), septic embolism, or unsecured aneurysm
3. Active bleeding
4. History of stroke in previous 6 weeks
5. Uncontrolled hypertension
6. Renal disease or renal dialysis
7. Treatment with any plasminogen activator within the last 48 hrs.
8. Therapy with a Glycoprotein IIb/IIIa inhibitor in 5 days prior to study enrollment or at any time during study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Saver, MD, Study Director — University of California, Los Angeles; Peter Mitchell, MD, Study Director — Melbourne Health
Locations (23):
- Australia (2):
  - Heidelberg Repatriation Hospital, Melbourne, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - Christian-Doppler-Klinik Salzburg,Universitätsklinik für Neurologie, Salzburg, Salzburg
  - O.O. Landes-Nervenklinik Wagner-Jauregg, Linz, Upper Austria
- France (4):
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Bichat-Claude Bernard, Paris
  - Hôpital Rangueil, Toulouse
- Serbia (5):
  - Clinical Center of Serbia, Clinic for Vascular and Endovascular Surgery, Belgrade
  - Special Hospital for Cerebrovascular Diseases "Sveti Sava", Belgrade
  - Clinical Center Kragujevac, Center for Radiology Diagnostic, Kragujevac
  - Clinical Center Niš, Center of Radiology, Niš
  - Clinical Center of Vojvodina, Center for Radiology, Novi Sad
- Slovakia (5):
  - Neurology Clinic Hospital with Policlinic of F.D. Roosevelt, Banská Bystrica
  - I. Neurology Clinic, University Hospital Bratislava, Bratislava
  - Radiology Clinic, University Hospital Martin, Martin
  - Neurology Clinic, Faculty Hospital Nitra, Nitra
  - Neurology Clinic, Central Military Faculty Hospital, Ružomberok
- Spain (5):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital General Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 20 mg Plasmin (Human) | 40 mg Plasmin (Human) | 80 mg Plasmin (Human)
Started | 8 | 16 | 16
Completed | 4 | 13 | 10
Not Completed | 4 | 3 | 6
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Death | 3 | 3 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population includes all subject who received any amount of Plasmin.
Groups:
- Safety Population: Plasmin (Human): Plasmin (Human), 20 mg, 40 mg, or 80 mg, delivered through a catheter into a thrombus
Arm/Group | Safety Population
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Region of Enrollment [Number; unit: participants]
  Serbia | 10
  France | 7
  Slovakia | 5
  Spain | 8
  Austria | 1
  Australia | 5
  Germany | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Symptomatic Intracranial Hemorrhage (SICH) by Dose Cohort
Time Frame: 90 days
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | 20 mg Plasmin (Human) | 40 mg Plasmin (Human) | 80 mg Plasmin (Human)
Number analyzed (Participants) | 8 | 16 | 16
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing the informed consent form up to the last day of the study, including the follow-up and off-study medication period, 90 days after treatment.
Description: Treatment-emergent adverse events were adverse events reported after the subject received study medication.
Arm/Group | 20 mg Plasmin (Human) | 40 mg Plasmin (Human) | 80 mg Plasmin (Human)
Serious Adverse Events (participants affected / at risk) | 6/8 | 7/16 | 7/16
Other Adverse Events (participants affected / at risk) | 8/8 | 12/16 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20 mg Plasmin (Human) (N=8) | 40 mg Plasmin (Human) (N=16) | 80 mg Plasmin (Human) (N=16)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Vascular disorders) | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 20 mg Plasmin (Human) (N=8) | 40 mg Plasmin (Human) (N=16) | 80 mg Plasmin (Human) (N=16)
HEADACHE (Nervous system disorders) | 2 | 2 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 1 | 0
MUSCLE SPASTICITY (Nervous system disorders) | 1 | 0 | 1
CENTRAL PAIN SYNDROME (Nervous system disorders) | 0 | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1 | 0
COMPLEX REGIONAL PAIN SYNDROME (Nervous system disorders) | 0 | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 0 | 1
HAEMORRHAGIC CEREBRAL INFARCTION (Nervous system disorders) | 0 | 0 | 1
HYPERTONIA (Nervous system disorders) | 0 | 0 | 1
NEURALGIA (Nervous system disorders) | 1 | 0 | 0
VASCULAR DEMENTIA (Nervous system disorders) | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 5 | 1 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 0 | 2
DIARRHOEA (Gastrointestinal disorders) | 0 | 2 | 0
FAECAL INCONTINENCE (Gastrointestinal disorders) | 2 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 0 | 1
MELAENA (Gastrointestinal disorders) | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 2 | 1
BRADYCARDIA (Cardiac disorders) | 0 | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0
PYREXIA (General disorders) | 3 | 2 | 5
OEDEMA PERIPHERAL (General disorders) | 1 | 2 | 0
CHEST PAIN (General disorders) | 1 | 0 | 1
DRUG INTOLERANCE (General disorders) | 0 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 2 | 1 | 3
BRONCHITIS (Infections and infestations) | 1 | 0 | 1
ORAL CANDIDIASIS (Infections and infestations) | 2 | 0 | 0
ABSCESS ORAL (Infections and infestations) | 0 | 0 | 1
BACTERAEMIA (Infections and infestations) | 0 | 0 | 1
BACTERIAL INFECTION (Infections and infestations) | 1 | 0 | 0
CANDIDIASIS (Infections and infestations) | 1 | 0 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 1 | 0 | 0
INFECTION (Infections and infestations) | 0 | 1 | 0
KERATITIS HERPETIC (Infections and infestations) | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
ORCHITIS (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
SEPSIS (Infections and infestations) | 0 | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 3 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 0
ANOREXIA (Metabolism and nutrition disorders) | 0 | 2 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0 | 1
CEREBRAL SALT-WASTING SYNDROME (Metabolism and nutrition disorders) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 1 | 1 | 1
INSOMNIA (Psychiatric disorders) | 2 | 0 | 1
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 | 2 | 0
AGITATION (Psychiatric disorders) | 0 | 1 | 1
DYSSOMNIA (Psychiatric disorders) | 0 | 0 | 2
SLEEP DISORDER (Psychiatric disorders) | 1 | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0 | 0
HALLUCINATION (Psychiatric disorders) | 1 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 1 | 2
HAEMATOMA (Vascular disorders) | 0 | 1 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 | 0 | 1
PHLEBITIS (Vascular disorders) | 0 | 1 | 0
THROMBOPHLEBITIS (Vascular disorders) | 0 | 0 | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 1 | 1
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 0 | 1
BLOOD GLUCOSE ABNORMAL (Investigations) | 1 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 2 | 1
EXCORIATION (Injury, poisoning and procedural complications) | 2 | 0 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 2 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 2 | 0 | 0
BLADDER DISTENSION (Renal and urinary disorders) | 1 | 0 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 1 | 0
INTERTRIGO (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the study, after providing sponsor 30 days' notice prior to submitting a manuscript or other materials related to the study to any outside party. At sponsor's request, site will remove any confidential information (other than study results), and site will upon sponsor's request delay publication or presentation for a period of up to 120 days to allow sponsor to protect its interests in any sponsor inventions.